CLINICAL TRIAL: NCT04636697
Title: Randomized, Observer-Blind, Placebo-Controlled, Phase 2/3 Study to Assess the Safety, Efficacy, and Immunogenicity of a Recombinant Coronavirus-Like Particle COVID-19 Vaccine in Adults 18 Years of Age or Older
Brief Title: Study of a Recombinant Coronavirus-Like Particle COVID-19 Vaccine in Adults
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-PRO-CoVLP-021; NCT04662697 (obsolete NCT alias)
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Injections, Intramuscular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (0.5 mL)
  Interventions: Drug: Intramuscular injection
- 3.75 µg of CoVLP Vaccine adjuvanted (Experimental): 3.75 µg of CoVLP adjuvanted vaccine with AS03 adjuvant (0.5 mL)
  Interventions: Biological: Intramuscular vaccine

INTERVENTIONS:
Drug: Intramuscular injection — Subjects will receive two doses of placebo given 21 days apart into the deltoid region of the alternating arm (each arm will be injected once)
  Arms: Placebo
Biological: Intramuscular vaccine — Subjects will receive two doses of 3.75 µg of CoVLP adjuvanted with AS03 adjuvant given 21 days apart into the deltoid region of the alternating arm (each arm will be injected once)
  Arms: 3.75 µg of CoVLP Vaccine adjuvanted

SUMMARY:
This Phase 2/3 study is a multi-portion design to confirm that the chosen formulation and dosing regimen of CoVLP has an acceptable immunogenicity and safety profile.

The Phase 3 portion is an event-driven, randomized, observer blinded, placebo-controlled design that will evaluate the efficacy and safety of the CoVLP formulation compared to placebo.

Subjects will be followed for safety and immunogenicity for a period of 12 months after the last vaccination.

ELIGIBILITY:
Inclusion criteria:

1. Subjects must have read, understood, and signed the informed consent form (ICF) prior to participating in the study; subjects must also complete study-related procedures and the subjects must communicate with the study staff at visits and by phone during the study;
2. At the Screening visit (Visit 1), male and female subjects must be:

   * Study Populations #1: 18 to 64 (has not yet had his/her 65th birthday) years of age, inclusive;
   * Study Population #2: 65 years of age or older;
   * Study Population #3: 18 years of age or older;
3. At Screening (Visit 1) and Vaccination (Visit 2), subject must have a body mass index (BMI) of:

   • Study Populations #1 and #2: ≥ 18.5 and < 30 kg/m2;
4. Subjects are considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study;
5. Study Population #1: Subjects must be in good general health prior to study participation, with no clinically relevant abnormalities that could jeopardize subject safety or interfere with study assessments, as determined by medical history, physical examination, and vital signs. Investigator discretion will be permitted with this inclusion criterion;

   All regions except Canada: Note: Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable and, according to the Investigator's judgment that must be documented in the source documents, the condition is unlikely to confound the results of the study or pose additional risk to the subject by participating in the study. Stable disease is generally defined as no new onset or exacerbation of pre-existing chronic disease three months prior to vaccination. Based on the Investigator's judgment, a subject with more recent stabilization of a disease could also be eligible.
6. Study Populations #1 and #3: Female subjects of childbearing potential must have a negative serum pregnancy test result at Screening (Visit 1 for the Phase 2 portion) and/or a negative urine pregnancy test result at Vaccination (Visit 2 for the Phase 2 portion; Visit 1 for the Phase 3 portion):

   Non-childbearing females are defined as:
   * Surgically-sterile (defined as bilateral tubal ligation, hysterectomy or bilateral oophorectomy performed more than one month prior to the first study vaccination); or
   * Post-menopausal (absence of menses for 12 consecutive months and age consistent with natural cessation of ovulation);
7. Study Populations #1 and #3: Female subjects of childbearing potential must use an effective method of contraception for one month prior to vaccination (Visit 2) and agree to continue employing highly effective birth control measures for at least one month after the last study vaccination (or in the case of early termination, she must not plan to become pregnant for at least one month after her last study vaccination).

   The following relationship or methods of contraception are considered to be highly effective:
   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
   * Oral;
   * Intravaginal;
   * Transdermal;
   * Progestogen-only hormonal contraception associated with inhibition of ovulation:
   * Oral;
   * Injectable;
   * Implantable;
   * Intra-uterine device with or without hormonal release;
   * Credible self-reported history of heterosexual vaginal intercourse abstinence prior to and for at least one month after the last study vaccination. Abstinent subjects who are ovulating should be asked what method(s) they would use should their circumstances change, and subjects without a well-defined plan should be excluded;
   * Female partner;
   * All regions except the US: Vasectomised partner, provided that this partner is the sole sexual partner of the study participant and that the vasectomised partner has received a medical assessment of the surgical success;
   * Bilateral tubal ligation.
8. Study Population #2: Subjects must be non-institutionalized (e.g. not living in rehabilitation centres or old-age homes; living in an elderly community is acceptable) and have no acute or evolving medical problems prior to study participation and no clinically relevant abnormalities that could jeopardize subject safety or interfere with study assessments, as assessed by the Principal Investigator or sub-Investigator (thereafter referred as Investigator) and determined by medical history, physical examination, serology (only for the Phase 2 portion), clinical chemistry and haematology tests (only for the Phase 2 portion), urinalysis (only for the Phase 2 portion), and vital signs. Investigator discretion will be permitted with this inclusion criterion.

   All regions except Canada: Note: Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable and, according to the Investigator's judgment that must be documented in the source documents, the condition is unlikely to confound the results of the study or pose additional risk to the subject by participating in the study. Stable disease is generally defined as no new onset or exacerbation of pre-existing chronic disease three months prior to vaccination. Based on the Investigator's judgment and documented in source documentation, a subject with more recent stabilization of a disease could also be eligible;
9. Study Population #3: Subjects must have one or more co-morbid conditions that puts them at higher risk for severe COVID-19 disease. These comorbidities include but are not limited to obesity, hypertension, type 1 or type 2 diabetes, chronic obstructive pulmonary disease (COPD), cardiovascular diseases, chronic kidney diseases, or be immunocompromised persons (e.g., treatment-controlled HIV infection, organ transplant recipients, or patients receiving cancer chemotherapy). Investigator discretion will be permitted with this inclusion criterion.

Exclusion criteria:

1. Study Populations #1 and #2: According to the Investigator's opinion, significant acute or chronic, uncontrolled medical or neuropsychiatric illness.

   Acute disease is defined as presence of any moderate or severe acute illness with or without a fever within 48 hours prior to the Screening (Visit 1) and/or Vaccination visit (Visit 2). 'Uncontrolled' is defined as:
   * Requiring a new medical or surgical treatment during the three months prior to study vaccine administration;
   * Requiring any significant change in a chronic medication (i.e. drug, dose, frequency) during the three months prior to study vaccine administration due to uncontrolled symptoms or drug toxicity unless the innocuous nature of the medication change meets the criteria outlined in inclusion criterion no. 5 (Study Population #1) or no. 8 (Study Population #2) and is appropriately justified and documented by the Investigator.

   Investigator discretion is permitted with this exclusion criterion and must be carefully and fully documented in the source documents;
2. Study Populations #1 and #2: Any chronic medical condition associated with elevated risk of severe outcomes of COVID-19, including obesity, diabetes (type 1 or type 2), significant cardiovascular or respiratory diseases including asthma, chronic renal failure, disorders of bleeding/coagulation, chronic inflammatory or autoimmune conditions, immunosuppressive conditions (including HIV), and hypertension;
3. Study Populations #1 and #2: Any confirmed or suspected current immunosuppressive condition or immunodeficiency, including cancer, human immunodeficiency virus (HIV), hepatitis B or C infection (subjects with a history of cured hepatitis B or C infection without any signs of immunodeficiency at present time are allowed). Investigator discretion is permitted with this exclusion criterion;
4. Study Populations #1 and #2: Current autoimmune disease (such as rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis or narcolepsy). Investigator discretion is permitted with this exclusion criterion, and subjects may be eligible to participate with appropriate written justification in the source document (i.e. subjects with a history of autoimmune disease who are disease-free without treatment for three years or more, or on stable thyroid replacement therapy, mild psoriasis [i.e. a small number of minor plaques requiring no systemic treatment], etc.);
5. Study Populations #1 and #2: Administration of any medication or treatment that may alter the vaccine immune responses, such as:

   * Systemic glucocorticoids at a dose exceeding 10 mg of prednisone (or equivalent) per day for more than seven consecutive days or for 10 or more days in total, within one month prior to the Vaccination visit (Visit 2). Inhaled, nasal, ophthalmic, dermatological, and other topical glucocorticoids are permitted;
   * Cytotoxic, antineoplastic, or immunosuppressant drugs - within 36 months prior to Vaccination (Visit 2);
   * Any immunoglobulin preparations or blood products, blood transfusion - within 6 months prior to Vaccination (Visit 2);
6. Study Population #3: Acute disease defined as presence of any moderate or severe acute illness with or without a fever within 48 hours prior to the Screening (Visit 1) and/or Vaccination visit (Visit 2);
7. Administration of any vaccine within 14 days prior to Vaccination (Visit 2); planned administration of any vaccine during the study (up to Day 28 of the study). Immunization on an emergency basis during the study will be evaluated on case-by-case basis by the Investigator;
8. Administration of any other SARS-CoV-2 / COVID-19, or other experimental coronavirus vaccine at any time prior to or during the study;
9. History of virologically-confirmed COVID-19;
10. Use of any investigational or non-registered product within 30 days or 5 half-lives, whichever is longer, prior to Vaccination (Visit 2) or planned use during the study period. Subjects who are in a prolonged post-administration observation period of another investigational or marketed drug clinical study, for which there is no ongoing exposure to the investigational or marketed product and all scheduled on-site visits are completed, will be allowed to take part in this study, if all other eligibility criteria are met;
11. Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at injection site that may interfere with injection site reaction rating. Investigator discretion will be permitted with this exclusion criterion;
12. Use of any prescription antiviral drugs with the intention of COVID-19 prophylaxis, including those that are thought to be effective for prevention of COVID-19 but have not been licensed for this indication, within one month prior to Vaccination (Visit 2);
13. For the Phase 2 portion of the study only: Use of prophylactic medications (e.g. antihistamines [H1 receptor antagonists], nonsteroidal anti-inflammatory drugs [NSAIDs], systemic and topical glucocorticoids, non-opioid and opioid analgesics) within 24 hours prior to the Vaccination (Visit 2) to prevent or pre-empt symptoms due to vaccination;
14. History of a serious allergic response to any of the constituents of CoVLP including AS03;
15. History of a documented anaphylactic reactions to plants or plant components (including tobacco, fruits and nuts);
16. Personal or family history of narcolepsy;
17. Subjects with a history of Guillain-Barré Syndrome;
18. Study Populations #1 and #3: Any female subject who has a positive or doubtful pregnancy test result prior to vaccination or who is lactating;
19. Subjects identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study, or any employees of Medicago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30918 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Phase 2 portion: Immediate adverse event (AEs) | 30 minutes
  Percentage, intensity, and relationship to vaccination of immediate AEs
Phase 2 portion: Solicited local and systemic adverse events (AEs) | 7 days
  Percentage, intensity, and relationship to vaccination of solicited local and systemic AEs
Phase 2 portion: Unsolicited adverse events (AEs) | 21 days
  Percentage, intensity, and relationship of unsolicited AEs
Phase 2 portion: Number of subjects with normal and abnormal clinically significant urine values | 3 days
  Number of subjects with normal and abnormal clinically significant urine values
Phase 2 portion: Number of subjects with normal and abnormal clinically significant haematological values | 3 days
  Number of subjects with normal and abnormal clinically significant haematological values
Phase 2 portion: Number of subjects with normal and abnormal clinically significant biochemical values | 3 days
  Number of subjects with normal and abnormal clinically significant biochemical values
Phase 2 portion: Percentage of subjects with normal and abnormal clinically significant urine values | 3 days
  Percentage of subjects with normal and abnormal clinically significant urine values
Phase 2 portion: Percentage of subjects with normal and abnormal clinically significant haematological values | 3 days
  Percentage of subjects with normal and abnormal clinically significant haematological values
Phase 2 portion: Percentage of subjects with normal and abnormal clinically biochemical values | 3 days
  Percentage of subjects with normal and abnormal clinically biochemical values
Phase 2 portion: Serious adverse events (SAEs), adverse events (AEs) leading to withdrawal, adverse event of special interest (AESI) (including vaccine-enhanced disease) and deaths | 21 days
  Percentage of SAEs, MAAEs, AEs leading to withdrawal, AESIs (including VED), and deaths
Phase 2 portion: Neutralizing antibody (Nab assay) response | Day 21
  Nab response induced in each Study Population against the SARS-CoV-2 virus
Phase 2 portion: Neutralizing antibody (Nab assay) response | Day 42
  Nab response induced in each Study Population against the SARS-CoV-2 virus
Phase 2 portion:Specific Th1 cell-mediated immunity (CMI) response | Day 21
  Specific Th1 CMI response induced in each Study Population against the SARS-CoV-2 , as measured by IFN-γ ELISpot
Phase 2 portion:Specific Th1 cell-mediated immunity (CMI) response | Day 42
  Specific Th1 CMI response induced in each Study Population against the SARS-CoV-2 , as measured by IFN-γ ELISpot
Phase 3 portion: Laboratory-confirmed (virologic method) symptomatic SARS-CoV-2 infection | Day 28 and after
  First occurrence, in a subject, of laboratory-confirmed (virologic method) symptomatic SARS-CoV-2 infection

SECONDARY OUTCOMES:
Phase 2 portion: Solicited local and systemic AEs (populations 1 and 2) | 7 days
  Relative percentage of solicited local and systemic AEs following each vaccine administration between the healthy adults (Study Population #1) and the healthy elderly population (Study Population #2, each age strata);
Phase 2 portion: Solicited local and systemic AEs (populations 1, 2 and 3) | 7 days
  Relative percentage of solicited local and systemic AEs by intensity grades for seven days following each vaccine administration between the healthy adults (Study Population #1) and the healthy elderly adults (Study Population #2) combined and the adults with significant comorbidities (Study Population #3)
Phase 2 portion: Serious adverse events (SAEs), medically attended adverse events (MAAEs), adverse events (AEs) leading to withdrawal, adverse event of special interest (AESI) (including vaccine-enhanced disease) and deaths | Day 43 to 386
  Percentage of SAEs, MAAEs, AEs leading to withdrawal, AESIs (including VED), and deaths
Phase 3 portion: Immediate adverse event (AEs) | 30 minutes
  Percentage, intensity, and relationship to vaccination of immediate AEs
Phase 3 portion: Solicited local and systemic AEs | 7 days
  Percentage, intensity, and relationship to vaccination of solicited local and systemic AEs
Phase 3 portion: Unsolicited adverse events (AEs) | 21 days
  Percentage, intensity, and relationship of unsolicited AEs
Phase 3 portion: Serious adverse events (SAEs), adverse events (AEs) leading to withdrawal, adverse event of special interest (AESI) (including vaccine-enhanced disease) and deaths | Day 0 to 386
  Percentage of SAEs, MAAEs, AEs leading to withdrawal, AESIs (including VED), and deaths
Phase 2 portion: Neutralizing antibody Geometric mean tiers (GMT) response (populations 1 and 2) | 21 days
  Relative neutralizing antibody response between the healthy adults (Study Population #1) and the healthy elderly population (Study Population #2; each age strata) will be analyzed using the Following parameter: Geometric mean tiers (GMT)
Phase 2 portion: Neutralizing antibody Geometric mean tiers (GMT) response (populations 1, 2 and 3) | 21 days
  • Relative neutralizing antibody response between the healthy adults (Study Population #1) and the healthy elderly adults (Study Population #2) combined and the adults with significant comorbidities (Study Population #3) will be analyzed using the Following parameter: Geometric mean tiers (GMT)
Phase 2 portion: Neutralizing antibody (Nab assay) response | Day 128
  Persistence of the Nab antibody response induced in each Study Population against the SARS-CoV-2 virus
Phase 2 portion: Neutralizing antibody (Nab assay) response | Day 201
  Persistence of the Nab antibody response induced in each Study Population against the SARS-CoV-2 virus
Phase 2 portion: Neutralizing antibody (Nab assay) response | Day 386
  Persistence of the Nab antibody response induced in each Study Population against the SARS-CoV-2 virus
Phase 2 portion: Specific antibody (IgG) response | Day 128
  Specific antibody response induced in each Study Population against the SARS-CoV-2 virus will be measured by the total IgG levels
Phase 2 portion: Specific antibody (IgG) response | Day 201
  Specific antibody response induced in each Study Population against the SARS-CoV-2 virus will be measured by the total IgG levels
Phase 2 portion: Specific antibody (IgG) response | Day 386
  Specific antibody response induced in each Study Population against the SARS-CoV-2 virus will be measured by the total IgG levels
Phase 2 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 21
  The ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 2 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 42
  The ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 2 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 128
  The ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 2 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 201
  The ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 2 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 386
  The ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 2 portion: Specific Th1 cell-mediated immunity (CMI) response | Day 201
  Specific Th1 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IFN-γ ELISpot
Phase 2 portion: Specific Th1 cell-mediated immunity (CMI) response | Day 386
  Specific Th1 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IFN-γ ELISpot
Phase 2 portion: Specific Th2 cell-mediated immunity (CMI) response | Day 21
  Specific Th2 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IL-4 (ELISpot)
Phase 2 portion: Specific Th2 cell-mediated immunity (CMI) response | Day 42
  Specific Th2 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IL-4 (ELISpot)
Phase 2 portion: Specific Th2 cell-mediated immunity (CMI) response | Day 201
  Specific Th2 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IL-4 (ELISpot)
Phase 2 portion: Specific Th2 cell-mediated immunity (CMI) response | Day 386
  Specific Th2 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IL-4 (ELISpot)
Phase 3 portion: Neutralizing antibody Geometric mean titers (GMT) response | Day 21
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Geometric mean titers (GMT)
Phase 3 portion: Neutralizing antibody Seroconversion (SC) rate response | Day 21
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Seroconversion (SC) rate
Phase 3 portion: Neutralizing antibody Geometric mean fold rise (GMFR) response | Day 21
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Geometric mean fold rise (GMFR)
Phase 3 portion: Neutralizing antibody Geometric mean titers (GMT) response | Day 42
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Geometric mean titers (GMT)
Phase 3 portion: Neutralizing antibody Seroconversion (SC) rate response | Day 42
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Seroconversion (SC) rate
Phase 3 portion: Neutralizing antibody Geometric mean fold rise (GMFR) response | Day 42
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Geometric mean fold rise (GMFR)
Phase 3 portion: Neutralizing antibody Geometric mean fold rise (GMFR) response | Day 201
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Geometric mean fold rise (GMFR)
Phase 3 portion: Neutralizing antibody Geometric mean titers (GMT) | Day 201
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Geometric mean titers (GMT)
Phase 3 portion: Neutralizing antibody Seroconversion (SC) rate response | Day 201
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Seroconversion (SC) rate
Phase 3 portion: Neutralizing antibody Geometric mean fold rise (GMFR) response | Day 386
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Geometric mean fold rise (GMFR)
Phase 3 portion: Neutralizing antibody Geometric mean titers (GMT) response | Day 386
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Geometric mean titers (GMT)
Phase 3 portion: Neutralizing antibody Seroconversion (SC) rate response | Day 386
  In a subset of subjects, Nab antibody response induced in each Study Population against the SARS-CoV-2 virus analyzed, using the following parameters: Seroconversion (SC) rate
Phase 3 portion: Specific antibody (IgG) response | Day 21
  In a subset of subjects, specific antibody response induced in each Study Population against the SARS-CoV-2 virus measured by the total IgG levels
Phase 3 portion: Specific antibody (IgG) response | Day 42
  In a subset of subjects, specific antibody response induced in each Study Population against the SARS-CoV-2 virus measured by the total IgG levels
Phase 3 portion: Specific antibody (IgG) response | Day 201
  In a subset of subjects, specific antibody response induced in each Study Population against the SARS-CoV-2 virus measured by the total IgG levels
Phase 3 portion: Specific antibody (IgG) response | Day 386
  In a subset of subjects, specific antibody response induced in each Study Population against the SARS-CoV-2 virus measured by the total IgG levels
Phase 3 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 21
  In a subset of subjects, the ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 3 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 42
  In a subset of subjects, the ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 3 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 201
  In a subset of subjects, the ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 3 portion: Neutralizing antibody titers: IgG ELISA antibody titers | Day 386
  In a subset of subjects, the ratio of neutralizing antibody titers:IgG ELISA antibody titers
Phase 3 portion: Specific Th1 cell-mediated immunity (CMI) response | Day 21
  In a subset of subjects, specific Th1 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IFN-γ ELISpot
Phase 3 portion: Specific Th1 cell-mediated immunity (CMI) response | Day 42
  In a subset of subjects, specific Th1 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IFN-γ ELISpot
Phase 3 portion: Specific Th1 cell-mediated immunity (CMI) response | Day 201
  In a subset of subjects, specific Th1 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IFN-γ ELISpot
Phase 3 portion: Specific Th1 cell-mediated immunity (CMI) response | Day 386
  In a subset of subjects, specific Th1 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IFN-γ ELISpot
Phase 3 portion: Specific Th2 cell-mediated immunity (CMI) response | Day 21
  In a subset of subjects, specific Th2 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IL-4 (ELISpot)
Phase 3 portion: Specific Th2 cell-mediated immunity (CMI) response | Day 42
  In a subset of subjects, specific Th2 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IL-4 (ELISpot)
Phase 3 portion: Specific Th2 cell-mediated immunity (CMI) response | Day 201
  In a subset of subjects, specific Th2 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IL-4 (ELISpot)
Phase 3 portion: Specific Th2 cell-mediated immunity (CMI) response | Day 386
  In a subset of subjects, specific Th2 CMI response induced in each Study Population against the SARS-CoV-2 virus; as measured by IL-4 (ELISpot)
Phase 2 portion: Laboratory-confirmed (virologic method) symptomatic SARS-CoV-2 infection | Day 28 to 386
  First occurrence, in a subject, of laboratory-confirmed (virologic method) symptomatic SARS-CoV-2 infection
Phase 2 portion: Severe COVID-19 disease | Day 28 to 386
  Percentage of severe COVID-19 disease
Phase 3 portion: Severe COVID-19 disease | Day 28 to 386
  Percentage of severe COVID-19 disease
Phase 3 portion: COVID-19-related symptoms in virologically-confirmed cases | through efficacy analysis, approximately 4 months
  Percentage and intensity of COVID-19-related symptoms
Phase 3 portion: Laboratory-confirmed asymptomatic SARS-CoV-2 infection | Day 201
  Percentage of laboratory-confirmed asymptomatic SARS-CoV-2 infection: confirmed by the ELISA method for the N protein
Phase 3 portion: Laboratory-confirmed symptomatic SARS-CoV-2 infection | through efficacy analysis, approximately 4 months
  First occurence, in a subject, of laboratory-confirmed symptomatic SARS-CoV-2 infection: virologic method
Phase 3 portion: Laboratory-confirmed symptomatic SARS-CoV-2 infection | Day 0 to 21
  First occurence, in a subject, of laboratory-confirmed symptomatic SARS-CoV-2 infection: virologic method
Phase 3 portion: Laboratory-confirmed symptomatic SARS-CoV-2 infection | Day 21 to 28
  First occurence, in a subject, of laboratory-confirmed symptomatic SARS-CoV-2 infection: virologic method
Phase 3 portion: Viral shedding after SARS-CoV-2 infection | through efficacy analysis, approximately 4 months
  Duration and intensity of viral shedding after SARS-CoV-2 infection
Phase 3 portion: Laboratory-confirmed symptomatic SARS-CoV-2 infection (by strain) | through efficacy analysis, approximately 4 months
  First occurrence, in a subject, of laboratory-confirmed symptomatic SARS-CoV-2 infection by strain: virologic method

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ward, MD, Study Director — Medicago
Locations (91):
- United States (45):
  - Achieve Clinical Research, LLC dba Accel Research Sites, Birmingham, Alabama
  - Fiel Family and Sports Medicine/CCT, Tempe, Arizona
  - Hope Clinical Research, Canoga Park, California
  - CNS Network, Garden Grove, California
  - Long Beach Clinical Trial Services Inc., Long Beach, California
  - Pharmacology Research Institute, Newport Beach, California
  - Wr-McCr, Llc, San Diego, California
  - Ascension Providence Health System, Washington D.C., District of Columbia
  - Alliance for Multispecialty Research, Coral Gables, Florida
  - Research Centers of America, Hollywood, Florida
  - AppleMed Research Inc, Miami, Florida
  - Elixia COVID-19, Palm Beach, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - ASR, LLC, Nampa, Idaho
  - Affinity Health, Chicago, Illinois
  - Meridian Clinical Research, Sioux City, Iowa
  - Benchmark Research, Covington, Louisiana
  - Ascension St. John Vaccine Research Unit, Grosse Pointe Woods, Michigan
  - Methodist Physicians, Fremont, Nebraska
  - Be Well Clinical Studies, LLC, Lincoln, Nebraska
  - Meridian Clinical Research LLC, Norfolk, Nebraska
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - Forte Family Practice/ CCT Research, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Meridian Clinical Research, Endwell, New York
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Trial Management Associates LLC, Wilmington, North Carolina
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Velocity Clinical Research Providence, Warwick, Rhode Island
  - Benchmark Research, Austin, Texas
  - Tekton Research, Austin, Texas
  - Global Medical Research, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Research Your Health, Plano, Texas
  - Mt. Olympus Medical Research, LLC, Sugar Land, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - DM Clinical Research/Martin Diagnostic Clinic, Tomball, Texas
  - South Ogden Family Medicine, Ogden, Utah
  - Advanced Clinical Research, Inc., West Jordan, Utah
- Argentina (5):
  - Mautalen Salud e Investigación (Expertia SA), Buenos Aires
  - Fundación FunDaMos, Buenos Aires
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Buenos Aires
  - Sanatorio Allende, Córdoba
  - Clinica Mayo de UMCB SRL, San Miguel de Tucumán
- Brazil (7):
  - Instituto de Pesquisas Clinicas L2IP, Brasília
  - Unidade Hospital do Rocio, Campo Largo
  - Santa Casa De Misericordia De Belo Horizonte, Minas Gerais
  - Centro de Pesquisa Clinica - Hospital Moinhos de Vento, Porto Alegre
  - IBPClin Instituto Brasil de Pequisa Clinica, Rio de Janeiro
  - Fundação Faculdade Regional de Medicina de Sao Jose do Rio Preto, São Paulo
  - Azidus Brasil Pesquisa e Desenvolvimento Ltda, Valinhos
- Canada (15):
  - CARe Clinic, Red Deer, Alberta
  - IWK Health Centre- Dalhousie University-Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - Dawson Clinical Research Inc., Guelph, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - LMC Clinical Research Inc. (CPU), Toronto, Ontario
  - Manna Research Toronto, Toronto, Ontario
  - Manna Research (Quebec), Lévis, Quebec
  - Manna Research (Mirabel), Mirabel, Quebec
  - McGill University Health Centre Vaccine Study Centre, Pierrefonds, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - Diex Research Quebec Inc., Québec, Quebec
  - Diex Recherche Joliette, Saint-Charles-Borromée, Quebec
  - Q&T Research Sherbrooke Inc., Sherbrooke, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
- Mexico (7):
  - Investigación Biomédica para el Desarrollo de Fármacos, S.A. de C.V., Aguascalientes
  - Centro para el Desarrollo de la Medicina y de Asistencia Médica Especializada S.C., Culiacán
  - RM Pharma Specialists S.A. de C.V., Mexico City
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigación Clínica en Yucatan S.C.P. (CEMDEICY S.C.P.), Mérida
  - Integra RGH Centro de Investigacion, Clinica de Ozonoterapia RGH AC, Puebla City
  - Sociedad de Metabolismo y Corazon S.C (SOMECO), Veracruz
  - Investigación Biomédica para el Desarrollo de Fármacos, S.A. de C.V., Zapopan
- United Kingdom (12):
  - NHS Grampian, Aberdeen
  - Synexus Midlands Clinical Research Centre, Birmingham
  - University Hospital Southampton NHS Foundation Trust (UHS), Bournemouth
  - Public Health Wales, Cardiff
  - Synexus Wales DRS, Cardiff
  - Mid and South Essex NHS Foundation Trust, Chelmsford
  - Synexus Lancashire DRS, Chorley
  - University Hospitals Derby and Burton, Derby
  - London North West University Healthcare NHS Trust, Harrow
  - Kings College Hospital, London
  - Synexus Manchester DRS, Manchester
  - University of York/York Teaching Hospital, York

REFERENCES:
- [Derived] Hager KJ, Perez Marc G, Gobeil P, Diaz RS, Heizer G, Llapur C, Makarkov AI, Vasconcellos E, Pillet S, Riera F, Saxena P, Geller Wolff P, Bhutada K, Wallace G, Aazami H, Jones CE, Polack FP, Ferrara L, Atkins J, Boulay I, Dhaliwall J, Charland N, Couture MMJ, Jiang-Wright J, Landry N, Lapointe S, Lorin A, Mahmood A, Moulton LH, Pahmer E, Parent J, Seguin A, Tran L, Breuer T, Ceregido MA, Koutsoukos M, Roman F, Namba J, D'Aoust MA, Trepanier S, Kimura Y, Ward BJ; CoVLP Study Team. Efficacy and Safety of a Recombinant Plant-Based Adjuvanted Covid-19 Vaccine. N Engl J Med. 2022 Jun 2;386(22):2084-2096. doi: 10.1056/NEJMoa2201300. Epub 2022 May 4. PMID 35507508
- See also: To obtain contact information for a study center near you, click here — https://covlpvaccine.com/